CLINICAL TRIAL: NCT02696460
Title: Efficacy of Inhaled 50% Equimolar Nitrous Oxide/Oxygen Gas Premix (Kalinox®) as Compared to Topically Administered 5% Eutectic Mixture of Lidocaine/Prilocaine (EMLA®) in Chronic Leg Ulcer Debridement
Brief Title: Efficacy of 50% Nitrous Oxide/50% Oxygen Gas Premix in Chronic Leg Ulcer Debridement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venenklinik Bellevue (Other)
Responsible Party: Principal Investigator, Juerg Traber, MD, Clinic Director Surgery, Venenklinik Bellevue
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VB_01_2010
Record Dates: First submitted 2015-12-08; First posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Leg Ulcer
Keywords: debridement; analgesia
MeSH Terms: conditions — Agnosia | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- N2O/O2 analgesia (Active Comparator): Wound debridement under analgesia with N2O/O2 premix.
  Interventions: Procedure: N2O/O2 analgesia; Procedure: Lidocaine/Prilocaine analgesia
- Lidocaine/Prilocaine analgesia (Active Comparator): Wound debridement under analgesia with eutectic mixture of 5% lidocaine/prilocaine.
  Interventions: Procedure: N2O/O2 analgesia; Procedure: Lidocaine/Prilocaine analgesia

INTERVENTIONS:
Procedure: N2O/O2 analgesia — Analgesia for ulcer debridement procedure is provided by the inhalation of N2O/O2 gas premix.
  Other Names: Kalinox® analgesia
Procedure: Lidocaine/Prilocaine analgesia — Analgesia for ulcer debridement procedure is provided by topically administered lidocaine/prilocaine cream.
  Other Names: EMLA® analgesia

SUMMARY:
Adequate analgesia in serial chronic leg ulcer debridement can be difficult to achieve. A common analgesia method is the topical administration of local anesthetics directly onto the wound. However, complete wound debridement is often hampered by insufficient analgesia leading to interruption of the actual debridement and fragmentation of treatment into more frequent serial debridement sessions. Alternatively, the inhalation of an nitrous oxide/oxygen (N2O/O2) gas premix could be used for analgesia. In this study, the investigators have compared the analgesic method of an eutectic mixture of topically administered lidocaine/prilocaine cream (EMLA®) with the inhalation of an equimolar 50% N2O/50% O2 gas premix (Kalinox®) in serial leg ulcer debridement.

DETAILED DESCRIPTION:
Study design: Prospective, controlled, single-center, cross-over design study. The study protocol was approved by the local ethical committee.

Study setting/participants: The study is performed in a highly specialized secondary care vein center. Patients with chronic foot and leg ulcer disease that are scheduled for repetitive ulcer debridement are eligible for the study and included into the study provided that written informed consent is obtained and no exclusion criteria are present.

Debridement procedure: For debridement, disposable sterile scalpel blades, ring curettes, and sterilized reusable scissors and forceps are used. The intended sharp mechanical debridement is proceeded as long as it is tolerated by the patient or terminated as planned. It will immediately be discontinued if the patient asks for it due to intolerable pain or discomfort.

Analgesia methods: For analgesia during debridement, either a topically administered eutectic mixture of 5% lidocaine/prilocaine (EMLA®) or an inhaled premix of 50% nitrous oxide/50% oxygen (Kalinox®) are used. The 5% lidocaine/prilocaine cream is administered as a thick layer directly onto the wound with a scoop and the wound is sealed with a polyurethane foil. After 30 minutes of exposure time, the foil is removed and debridement is started immediately. For analgesia with the inhaled 50% nitrous oxide/50% oxygen premix, the patient is asked to hold an inhalation rebreather mask with on-demand-valve tightly placed onto the face after being instructed on how to inhale the gas premix. After 3 minutes of exposure time to the gas premix, debridement is started immediately. Gas inhalation is sustained until final wound dressing is applied. During the entire procedure with each analgesia method, vital signs such as non-invasive blood pressure, heart rate and peripheral oxygen saturation (SpO2) are be recorded.

Allocation of the analgesia regimen: After study enrollment, patients are consecutively numbered starting at one. Even numbered patients have the first debridement done with topical administration of lidocaine/prilocaine cream, followed by inhaled nitrous oxide/oxygen premix for the second debridement, and again followed in an alternating way by both tested analgesia methods up to a maximum of 4 interventions. Uneven numbered patients receive inhaled nitrous oxide/oxygen premix first, followed by topical lidocaine/prilocaine cream. After 4 debridement in total with 2 sets of each analgesia method, the study period for each single patient will be secluded. A maximum of 4 data sets per patient will be brought to data analysis.

Outcome measures: Primary outcome is the change of pain perception from baseline (1 minute before debridement) to time point of maximum debridement/wound profoundness (up to 10 minutes after start of debridement) as measured by the visual analogue scale (VAS). Secondary outcomes are change of pain perception from time point of maximum debridement/wound profoundness to 5 minutes after debridement as measured by the visual analogue scale (VAS), duration of treatment session, duration of debridement, achievement of treatment goal (completion), subjective general perception of analgesia quality during debridement (patient comfort). Baseline characteristics are gender, age, ulcer etiology, time passed between initial ulcer diagnosis and first debridement, wound emergence in terms of suspected trigger for ulcer development, and wound size.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic leg ulcer persisting for more than six weeks despite initial conservative treatment; written informed consent

Exclusion Criteria:

* Other chronic wounds than leg ulcers
* Peripheral polyneuropathy
* Non-specified peripheral sensibility disorders
* Allergies or contraindications against the study agents
* Lack of informed consent
* Pregnancy or breast feeding
* Anticipated need for less than two surgical debridement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change of Pain Level as Measured by Visual Analogue Scale (VAS) | Change of VAS from Time Point "Baseline 1 Minute before Start of Surgical Debridement" at Time Point "End of Surgical Debridement up to 10 Minutes after Start of Surgical Debridement"
  Change of measured VAS between Time Point "Baseline", which is 1 Minute Before Start of Surgical Debridement, and Time Point "End of Surgical Debridement", which is at Maximum Wound Profoundness and up to 10 Minutes after Start of Surgical Debridement.

SECONDARY OUTCOMES:
Change of Pain Level as Measured by Visual Analogue Scale (VAS) | Change of VAS from Time Point "End of Surgical Debridement" at Time Point "5 Minutes After Surgical Debridement"
  Change of measured VAS between Time Point "End of Surgical Debridement", which is at Maximum Wound Profoundness during Debridement, and Time Point "5 Minutes after Surgical Debridement".
Overall Duration of Treatment Session | From Admission to Discharge up to 60 Minutes
  Time Patient Spent in Outpatient Clinic for Treatment Session
Duration of Wound Debridement | From Start to End of Debridement up to 10 Minutes
  Total Procedure Time of Debridement
Achievement of Treatment Goal | From Start to End of Debridement up to 10 Minutes
  Surgeon's Judgement whether Debridement was Completed as Planned or Interrupted Prematurely due to Pain and/or Patient Discomfort.
Overall Analgesia Quality | From Start to End of Debridement up to 10 Minutes
  Patient's Subjective Perception of Analgesia Quality within the Time Frame of Debridement.

CONTACTS AND LOCATIONS:
Overall Officials: Juerg Traber, MD, Principal Investigator — Venenklinik Bellevue

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauer C, Lahjibi-Paulet H, Somme D, Onody P, Saint Jean O, Gisselbrecht M. Tolerability of an equimolar mix of nitrous oxide and oxygen during painful procedures in very elderly patients. Drugs Aging. 2007;24(6):501-7. doi: 10.2165/00002512-200724060-00006. PMID 17571915
- [Background] Onody P, Gil P, Hennequin M. Safety of inhalation of a 50% nitrous oxide/oxygen premix: a prospective survey of 35 828 administrations. Drug Saf. 2006;29(7):633-40. doi: 10.2165/00002018-200629070-00008. PMID 16808555
- [Background] Zwakhalen SM, Hamers JP, Berger MP. Improving the clinical usefulness of a behavioural pain scale for older people with dementia. J Adv Nurs. 2007 Jun;58(5):493-502. doi: 10.1111/j.1365-2648.2007.04255.x. Epub 2007 Apr 17. PMID 17442027
- [Background] Annequin D, Carbajal R, Chauvin P, Gall O, Tourniaire B, Murat I. Fixed 50% nitrous oxide oxygen mixture for painful procedures: A French survey. Pediatrics. 2000 Apr;105(4):E47. doi: 10.1542/peds.105.4.e47. PMID 10742368
- [Background] Evans E, Gray M. Do topical analgesics reduce pain associated with wound dressing changes or debridement of chronic wounds? J Wound Ostomy Continence Nurs. 2005 Sep-Oct;32(5):287-90. doi: 10.1097/00152192-200509000-00002. No abstract available. PMID 16234718
- [Background] Hee HI, Goy RW, Ng AS. Effective reduction of anxiety and pain during venous cannulation in children: a comparison of analgesic efficacy conferred by nitrous oxide, EMLA and combination. Paediatr Anaesth. 2003 Mar;13(3):210-6. doi: 10.1046/j.1460-9592.2003.01051.x. PMID 12641682
- [Background] Doughty DB. Strategies for minimizing chronic wound pain. Adv Skin Wound Care. 2006 Mar;19(2):82-5. doi: 10.1097/00129334-200603000-00009. No abstract available. PMID 16557053
- [Background] Rosenthal D, Murphy F, Gottschalk R, Baxter M, Lycka B, Nevin K. Using a topical anaesthetic cream to reduce pain during sharp debridement of chronic leg ulcers. J Wound Care. 2001 Jan;10(1):503-5. doi: 10.12968/jowc.2001.10.1.26042. PMID 12964231
- [Background] Holm J, Andren B, Grafford K. Pain control in the surgical debridement of leg ulcers by the use of a topical lidocaine--prilocaine cream, EMLA. Acta Derm Venereol. 1990;70(2):132-6. PMID 1969197